CLINICAL TRIAL: NCT00682981
Title: A Phase I Followed by a Randomized, Phase II Study of Carboplatin and Etoposide With or Without Obatoclax Administered Every 3 Weeks to Patients With Extensive- Stage Small Cell Lung Cancer (ES-SCLC)
Brief Title: A Phase I/II Study of Carboplatin and Etoposide With or Without Obatoclax in Extensive-stage Small Cell Lung Cancer (ES-SCLC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gemin X (Industry)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEM017
Record Dates: First submitted 2008-05-20; First posted 2008-05-23 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Extensive-stage Small Cell Lung Cancer
Keywords: ES-SCLC; Obatoclax
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — obatoclax; EC regimen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Phase I A (Experimental): Obatoclax for 3 hours for 3 days with carboplatin/etoposide.
  Interventions: Drug: Obatoclax; Drug: Carboplatin/etoposide
- Phase I B (Experimental): Obatoclax for 24 hours for 3 days with carboplatin/etoposide.
  Interventions: Drug: Obatoclax; Drug: Carboplatin/etoposide
- Phase II A (Experimental): Obatoclax for 3 hours for 3 days with carboplatin/etoposide.
  Interventions: Drug: Obatoclax; Drug: Carboplatin/etoposide
- Phase II B (Active Comparator): Carboplatin/etoposide without continued study treatment
  Interventions: Drug: Carboplatin/etoposide

INTERVENTIONS:
Drug: Obatoclax — IV Infusions for 3 consecutive days of either 3-hours, 2 hours duration
  Other Names: GX15-070MS
  Arms: Phase I A; Phase I B; Phase II A
Drug: Carboplatin/etoposide — Carboplatin/etoposide combination
  Other Names: Control

SUMMARY:
The Phase I portion of this protocol will determine the best phase II dose and schedule of obatoclax with carboplatin and etoposide in patients with extensive-stage small cell lung cancer. The Phase II portion will evaluate the response rate to this regimen.

DETAILED DESCRIPTION:
In the Phase I portion, both 3 hour and 24 hour infusions of obatoclax with carboplatin and etoposide every 3 weeks will be evaluated at different doses. In the Phase II portion, 3 hour infusions of obatoclax with or without carboplatin and etoposide every three weeks will be evaluated for response rates.

ELIGIBILITY:
Inclusion Criteria:

Phase I:

* Pathological or cytological confirmation of SCLC
* ES-SCLC
* Measurable disease using Response Evaluation Criteria in Solid Tumors (RECIST) with at least one lesion ≥2.0 cm using conventional technique or ≥1.0 cm with spiral computed tomography (CT) scan in a single dimension
* No previous chemotherapy
* Age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1
* Normal organ function defined as: absolute neutrophil count (ANC)

  * 1500/mm3, platelets ≥100,000/mm3, total bilirubin ≤ upper limit of normal (ULN) or total bilirubin ≤ 3.0 if liver metastases are present, alanine aminotransferase (serum glutamic pyruvic transaminase) (ALT [SGPT])

    * 2.5 ´ ULN or ALT/SGPT ≤ 5 ´ ULN if liver metastases are present, and creatinine within normal institutional limits or calculated creatinine clearance ≥50 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Negative serum or urine pregnancy test result prior to study entry. In addition, women of child-bearing potential and men with partners of child-bearing potential must agree to use acceptable forms of birth control (those that result in less than 1% pregnancy/year when used correctly: implants, injectables, combined oral contraceptives, some IUDs, vasectomy of a male partner, sexual abstinence)
* Ability to understand and willingness to sign a written informed consent form

Phase II:

* Pathological or cytological confirmation of SCLC
* ES-SCLC
* Measurable disease using RECIST criteria with at least one lesion

  * 2.0 cm using conventional technique or ≥1.0 cm with spiral CT scan in a single dimension
* No previous chemotherapy
* Age ≥18 years
* ECOG Performance Status ≤2;
* Normal organ function defined as: ANC ≥1500/mm3, platelets ≥100,000/mm3, total bilirubin ≤ULN or total bilirubin ≤ 3.0 if liver metastases are present, ALT (SGPT) ≤2.5 ´ ULN or ALT/SGPT ≤ 5 ´ ULN if liver metastases are present, and creatinine within normal institutional limits or calculated creatinine clearance ≥50 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Negative serum or urine pregnancy test result prior to study entry. In addition, women of child-bearing potential and men with partners of child-bearing potential must agree to use acceptable forms of birth control (those that result in less than 1% pregnancy/year when used correctly: implants, injectables, combined oral contraceptives, some IUDs, vasectomy of a male partner, sexual abstinence)
* Ability to understand and willingness to sign a written informed consent form

Exclusion Criteria:

Phase I and II:

* Other investigational or commercial agents or therapies administered with the intent to treat the patient's malignancy
* History of allergic reactions attributed to components of the obatoclax formulation (Polysorbate 20 and PEG 300)
* History of seizure disorders unrelated to SCLC brain metastases, or presence of symptomatic brain metastases
* Uncontrolled,intercurrent illness including, but not limited to, symptomatic neurological illness; active, uncontrolled systemic infection considered opportunistic, lifethreatening,or clinically significant at the time of treatment; symptomatic congestive heart failure; unstable angina pectoris; clinically significant cardiac arrhythmia; significant pulmonary disease or hypoxia; or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women and women who are breast feeding;
* human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2008-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Determine the recommended Phase II dose of obatoclax administered as a 3-hour or 24-hour infusion for 3 consecutive days in Phase I, and response rate in Phase II. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean Viallet, MD, Study Director — Gemin X Pharmaceuticals
Locations (75):
- United States (32):
  - Clearview Cancer Institute, Huntsville, Alabama
  - Northwest Alabama Cancer Center, Muscle Shoals, Alabama
  - Mayo Clinic-Arizona, Scottsdale, Arizona
  - Arizona Clinical Research Center, Tucson, Arizona
  - City of Hope and Beckman Research Institute, Duarte, California
  - University of California-San Diego Moores Cancer Center, La Jolla, California
  - Georgetown University Hospital-Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Integrated Community Oncology Network, Jacksonville, Florida
  - University of Miami-Sylvester Cancer Center, Miami, Florida
  - Florida Cancer Institute, New Port Richey, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Northwest Georgia Oncology Centers, Marietta, Georgia
  - University of Chicago, Chicago, Illinois
  - Iowa Blood and Cancer Center, PLC, Cedar Rapids, Iowa
  - Cancer Center of Kansas, Wichita, Kansas
  - James Brown Cancer Center, Louisville, Kentucky
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Kalamazoo Hematology and Oncology, Kalamazoo, Michigan
  - Mid Ohio Oncology/Hematology, Inc., Columbus, Ohio
  - Cancer Care Associates-Oklahoma City, Oklahoma City, Oklahoma
  - Cancer Care Associates-Tulsa, Tulsa, Oklahoma
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - Greater Philadelphia Cancer and Hematology Specialists, Philadelphia, Pennsylvania
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - McLeod Cancer & Blood Center, Johnson City, Tennessee
  - The West Clinic, Memphis, Tennessee
  - Baylor, Dallas, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Peninsula Cancer Institute, Newport News, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Wheeling Hospital, Wheeling, West Virginia
- Bulgaria (4):
  - MHAT "Dr. Tota Venkova", Gabrovo
  - District Dispensary for Cancer Diseases, Plovdiv, Plovdiv
  - District Dispensary for Oncology Diseases, Sofia City, Sofia
  - Specialized Hospital for Active Treatment in Oncology, Sofia
- Canada (3):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - McGill University, Montreal, Quebec
- Czechia (5):
  - Regional Hospital Kladno, Kladno
  - Hospital Kutna Hora, Kutná Hora
  - University Hospital Olomouc, Olomouc
  - Faculty Hospital Ostrava, Ostrava-Poruba
  - University Hospital Na Bulovce, Prague
- Hungary (8):
  - National Institute of Tuberculosis & Pulmonology, Budapest
  - Semmelweis University Medical School, Budapest, Budapest
  - University Of Debrecen Medical and Health Science Centre, Debrecen
  - Csongrad County Council's Hospital for Chest Diseases, Deszk
  - Bacs-Kiskun County Hospital, Kecskemét
  - State Hospital Matrahaza, Mátraháza
  - Clinfan Ltd. SMO Tolna County Hospital, Szekszárd
  - Pest County Hospital, Törökbálint
- India (8):
  - Vedanta Institute of Medical Sciences, Ahmedabad, Gujarat
  - Kailash Cancer Hospital and Research Centre, Goraj, Gujarat
  - Jawaharlal Nehru Cancer Hospital and Research Centre, Bhopal, Madhya Pradesh
  - Curie Manavata Cancer Centre, Nashik, Maharashtra
  - Noble Hospital, Pune, Maharashtra
  - Dr. Kamakshi Memorial Hospital, Chennai, Tamal Nadu
  - Galaxy Cancer Institute, Pushpanjali Crosslay Hospital, Ghaziabad, Uttar Pradesh
  - Orchid Nursing Home, Kolkata, West Bengal
- Poland (5):
  - Wojewodzki Szpital Specjalistyczny im. K. Dluskiego, Bialystok
  - SPZ Gruzlicy i Chorob Pluc, Olsztyn
  - Mazowieckie Centrum Leczenia Chorob Pluc i Gruzlicy, Otwock
  - Specjalistyczny Szpital im Prof Alfreda Sokolowskiego, Szczecin-Zdunowo
  - Wojewodzki Szpital Chorob Pluc, Wodzisław Śląski
- Romania (3):
  - Prof. Dr. Ion Chiricuta Oncology Institute Cluj Napoca, Cluj-Napoca
  - Oncology Medical Centre SCM, Iași
  - Emergency Clinical County Hospital Oradea, Oradea
- Serbia (2):
  - Institute for Pulmonary Diseases of Vojvodina, Kamenitz
  - Center for Pulmonary Diseases, Clinic for Internal Medicine, Kragujevac
- United Kingdom (5):
  - Northern Ireland Cancer Centre Queens University Belfast, Belfast, Northern Ireland
  - Royal Bournemouth Hospital, Dorset
  - Nottingham University Hospital, Nottingham
  - Weston Park Hospital, Sheffield
  - Royal Surrey County Hospital, Surrey

REFERENCES:
- [Derived] Langer CJ, Albert I, Ross HJ, Kovacs P, Blakely LJ, Pajkos G, Somfay A, Zatloukal P, Kazarnowicz A, Moezi MM, Schreeder MT, Schnyder J, Ao-Baslock A, Pathak AK, Berger MS; GEM017 Investigators. Randomized phase II study of carboplatin and etoposide with or without obatoclax mesylate in extensive-stage small cell lung cancer. Lung Cancer. 2014 Sep;85(3):420-8. doi: 10.1016/j.lungcan.2014.05.003. Epub 2014 May 13. PMID 24997137